CLINICAL TRIAL: NCT03870750
Title: Seamless Phase II-Phase III Randomized Clinical Trial to Identify and Confirm the Most Promising Novel Intervention to Alleviate Morbidity and Mortality After Allogeneic Hematopoietic Cell Transplantation Among Older, Medically Infirm, or Frail Patients With Hematological Diseases
Brief Title: Identifying Best Approach in Improving Quality of Life and Survival After a Donor Stem Cell Transplant in Older, Medically Infirm, or Frail Patients With Blood Diseases
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study terminated due to meeting interim analysis futility endpoint. No difference was found between two treatment arms at interim analysis of primary outcome.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1004746; NCI-2019-01097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9885 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA227092 (NIH)
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Non-Neoplastic Hematologic and Lymphocytic Disorder
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Palliative Care; Patient Comfort; Practice Guidelines as Topic; Standard of Care; Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm I (SPC) (Experimental): Patients undergo SPC on days -15 before to +56 after transplant. Patients undergo HCT on day 0 and complete questionnaires and surveys at enrollment, 30, 90, 180, and 365 days post HCT. Patients complete a 4-meter walk test, 6-minute walk test, up and go test, measured strength test and cognitive assessment at enrollment, 90, 180, and 365 days post HCT. Patients may also complete surveys on medical and non-medical (transportation, lodging) costs related to transplant after HCT.
  Interventions: Other: Supportive Palliative Care; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Other: Survey Administration
- Arm II (CMC) (Experimental): Patients undergo a CMC program on days -15 to 56. Patients undergo HCT on day 0 and complete questionnaires and surveys at enrollment, 30, 90, 180, and 365 days post HCT. Patients complete a 4-meter walk test, 6-minute walk test, up and go test, measured strength test and cognitive assessment at enrollment, 90, 180, and 365 days post HCT. Patients may also complete surveys on medical and non-medical (transportation, lodging) costs related to transplant after HCT.
  Interventions: Other: Clinical Management; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Other: Survey Administration
- Arm III (SPC and CMC) (Experimental): Patients undergo interventions as outlined in Arm I and Arm II. Patients undergo HCT on day 0 and complete questionnaires and surveys at enrollment 30, 90, 180, and 365 days post HCT. Patients complete a 4-meter walk test, 6-minute walk test, up and go test, measured strength test and cognitive assessment at enrollment, 90, 180, and 365 days post HCT. Patients may also complete surveys on medical and non-medical (transportation, lodging) costs related to transplant after HCT.
  Interventions: Other: Supportive Palliative Care; Other: Clinical Management; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Other: Survey Administration
- Arm IV (standard of care) (Active Comparator): Patients receive standard of care. Patients undergo HCT on day 0 and complete questionnaires and surveys at enrollment, 30, 90, 180, and 365 days post HCT. Patients complete a 4-meter walk test, 6-minute walk test, up and go test, measured strength test and cognitive assessment at enrollment, 90, 180, and 365 days post HCT. Patients may also complete surveys on medical and non-medical (transportation, lodging) costs related to transplant after HCT.
  Interventions: Other: Best Practice; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Other: Supportive Palliative Care — focuses on relieving symptoms of stress from serious illness and care through physical, cultural, psychological, social, spiritual, and ethical aspects
  Other Names: Comfort Care; palliation; palliative care; palliative therapy; Palliative Treatment; Symptom Management; Symptoms Management; PA-Palliative Therapy
  Arms: Arm I (SPC); Arm III (SPC and CMC)
Other: Clinical Management — physical exercise, strength training, stress reduction, medication management, dietary recommendations, and education
  Arms: Arm II (CMC); Arm III (SPC and CMC)
Other: Best Practice — Given standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm IV (standard of care)
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation
  Arms: Arm I (SPC); Arm II (CMC); Arm III (SPC and CMC)
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Complete surveys

SUMMARY:
This phase II/III trial studies the best approach in improving quality of life and survival after a donor stem cell transplant in older, weak, or frail patients with blood diseases. Patients who have undergone a transplant often experience increases in disease and death. One approach, supportive and palliative care (SPC), focuses on relieving symptoms of stress from serious illness and care through physical, cultural, psychological, social, spiritual, and ethical aspects. While a second approach, clinical management of comorbidities (CMC) focuses on managing multiple diseases, other than cancer, such as heart or lung diseases through physical exercise, strength training, stress reduction, medication management, dietary recommendations, and education. Giving SPC, CMC, or a combination of both may work better in improving quality of life and survival after a donor stem cell transplant compared to standard of care in patients with blood diseases.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 4 arms.

ARM I: Patients undergo SPC on days -15 before to +56 after transplant.

ARM II: Patients undergo a CMC program on days -15 before to +56 after transplant.

ARM III: Patients undergo interventions as outlined in Arm I and Arm II.

ARM IV: Patients receive standard of care.

In all arms, patients undergo HCT on day 0 and complete questionnaires and surveys at enrollment and 30, 90, 180, and 365 days post HCT. In all arms patients complete a 4-meter walk test, 6-minute walk test, up and go test, measured strength test and cognitive assessment at enrollment, 90, 180, and 365 days post HCT. Patients may also complete surveys on medical and non-medical (transportation, lodging) costs related to transplant after HCT.

ELIGIBILITY:
Inclusion Criteria:

* Vulnerable patients as defined by one or more of the following criteria

  * Age 65 years or older
  * Having Hematopoietic Cell Transplantation - Comorbidity Index (HCT-CI) scores of >= 3 (for patients that could be 20 years old and older)
  * Having frailty as determined by walk speed of < 0.8 m/s using 4-meter walk test (for patients 50 years old and older)
* Patients considered or referred for allogeneic HCT to treat a hematological malignant or non-malignant disease
* Able to speak and read English - interaction with the interventionist trainer and endpoint measurement must occur in English
* Willing and able to provide informed consent
* Planned allogeneic HCT within 3 weeks - all types of donors and all sorts of conditioning regimens are allowed. Patients with suspected active disease (relatively old disease staging or relatively old intervention) or significant comorbidity (e.g. suspicious untreated pulmonary nodules) based on prior evaluations, that could delay the transplant would be considered for enrollment within a tighter window (10-14 days before allogeneic HCT) to allow for completed pre-HCT work-up evaluations that would confirm readiness to proceed with transplant
* Able to exercise at low to moderate intensity, specifically taking into consideration the rare circumstances where subjects are not able to exercise due to either birth deformity or prior traumatic injury that affects their gait
* Adequate cardiopulmonary reserve, as judged by data from the patient's electronic medical record as to whether a patient could walk up one flight of stairs, no need for supplemental oxygen, and/or physician judgment

Exclusion Criteria:

* Orthopedic, neurologic or other problems which prevent safe ambulation and protocol adherence. Information on prior falls and other recent orthopedic or neurologic problems will be used to make judgment about protocol eligibility
* Participation in another intervention clinical trial with HRQOL as a primary endpoint
* Planned donor lymphocyte infusion (DLI) within 90 days post-transplant
* Planned anti-cytotoxic therapies, other than tyrosine kinase inhibitors or single-agent monoclonal antibody, or FLT-3 inhibitors within 90 days of post-transplant unless pre-approved by the protocol principal investigator (PI)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in health-related quality of life (HRQOL) (Phase II) | First 90 days after HCT
  The arm with the largest mean change in Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) from baseline to day 90. The Wilcoxon rank-sum test will be used to compare change in FACT-BMT between arms, and this will also be the test to be used in computation of the conditional power at the end of phase II.
Survival after hematopoietic cell transplantation (HCT) (Phase III) | At 1 year after HCT
Change in HRQOL (Phase III) | Baseline to 90 days post-HCT
  Will be measured by the FACT-BMT.

SECONDARY OUTCOMES:
Rate of overall survival | Up to 1 year
  Overall survival will be compared between each of the experimental arms and the usual care only (UCO) arm using the log-rank test. Arms that do not survive the screening phase will also be included for comparison.
Non-relapse mortality | At 90 days and up to 1 year
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; analysis of variance (ANOVA) or Kruskal-Wallis test for comparisons involving more than two groups). Will use generalized estimating equations (GEEs) approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Cumulative incidence of relapse | Up to 1 year
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Relapse-free survival | Up to 1 year
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Cumulative incidence of frailty | Up to 1 year
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Cumulative incidence of disability | Up to 1 year
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Frequency of hospitalization | Up to 90 days after HCT
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Duration of each hospitalization | Up to 90 days after HCT
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Number of admissions to intensive care unit | Up to 90 days after HCT
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Duration of admissions to intensive care unit | Up to 90 days after HCT
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.
Days out of hospital alive | Up to 90 days after HCT
  Will be compared between arms using appropriate tests for continuous data (two-sample t-test or Wilcoxon rank-sum test, as appropriate for two-group comparisons; ANOVA or Kruskal-Wallis test for comparisons involving more than two groups). Will use GEEs approach for regression models, which can accommodate the within patient correlation structure and arbitrary patterns of missing data and also allow for the population average interpretation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sorror, MD, MSc, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (11):
- United States (11):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health Cancer Institute, New Hyde Park, New York
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT03870750/ICF_000.pdf